CLINICAL TRIAL: NCT01462071
Title: Red Blood Cell Lifespan and Inflammation in Dialysis Patients
Brief Title: Red Blood Cell Lifespan
Acronym: RBC
Status: Terminated | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 039-08
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Kidney Disease; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease

SUMMARY:
Background:

A low amount of red blood cells in the blood of patients with limited kidney function is a well known problem. Besides the lack of substances in the blood like iron or erythropoietin the shortened survival of red blood cells leads to the low red blood cell count. Red blood cells of patients on kidney replacement therapy (dialysis) die earlier than those of healthy persons. They live only about 70 days compared to 120 days in healthy humans. Today little is known about the causes for the shorter survival of the red blood cells in patients on dialysis. Because inflammation leads to a shorter life of the red blood cells in people suffering from several diseases leading to inflammation we would like to learn about the role of inflammation in the shortened life of red blood cells of dialysis patients.

When red blood cells are dying the content is broken down to several substances. One of these substances is the gas carbon monoxide (CO). The carbon monoxide is exhaled with the breath. The more red blood cells die the more CO is exhaled. That's why we can calculate the lifespan of the red blood cells when we measure the amount of CO in breath at the same time as the red blood cell count in the blood.

Aim of the study:

We aim to learn about the influence of inflammation of on red blood cell survival in dialysis patients. To look for factors with effect on inflammation or red blood cell survival, for example type of dialysis access, medication or kind of dialysis treatment.

Study procedures:

Over the course of the 18 month study, 6 observational assessments will take place. If the patient experiences a situation with increased inflammation during the study period (for example any kind of infection or intervention) up to two more study visits will take place. Each study visit will include blood sampling, performed without the need for an extra needle stick, and a breath sampling in order to calculate the red blood survival and to measure markers for inflammation in the blood. The breath sample will be taken using the easy to use GaSampler device developed by a company called Quintron especially for medical breath sampling.

In order to get a sample of air at the patient's home for calculation of carbon monoxide produced in the body we will ask the patients to take home an open empty plastic bottle before each study visit. The bottle should be kept overnight on a table or sideboard in the apartment. Before leaving home for hemodialysis or in clinic visit the patient will seal the plastic bottle with the top, take it to the dialysis center and hand it to the research staff.

Risks:

The amount of the additional blood drawn is 30 ml; this is the amount 2 tablespoons, at each study visit. This does not harm the patient. The breath sampling does not imply any risk.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Chronic hemo- or peritoneal dialysis treatment greater than 3 months

Exclusion Criteria:

* Inability to understand the English language and give informed consent for participation in the study

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult patients (at least 18 years of age) who perform chronic peritoneal dialysis treatment or hemodialysis treatment. Both men and women can participate in the study, and no race or ethnic group will be excluded. No subjects that require special protections will be involved.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Relationship between inflammation and erythrocyte lifespan | 6 visits during 18 month period

SECONDARY OUTCOMES:
Evaluate the accuracy of HbA1c and fructosamine measurements for assessment of glucose control | 6 visits during 18 month period

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Yorkville Dialysis Center, New York, New York, United States